CLINICAL TRIAL: NCT01529801
Title: A Prospective Randomized-controlled Study of the Effect of Surface Topographies on Implant Integration Rates and Clinical Success
Brief Title: Assessment of the Effect of a Novel Surface Roughness Treatment on Dental Implants on Integration Success
Acronym: Luna
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3011
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: edentulism; dental implants; clinical study; randomized; Osseotite Certain Tapered; Crestal bone level
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Roughness group A (Experimental): Osseotite Certain Tapered Group A
  Interventions: Device: Osseotite Certain Tapered Group A
- Roughness Group B (Experimental): Osseotite Certain Tapered Group B
  Interventions: Device: Osseotite Certain Tapered Group B
- Roughness Group C (Experimental): Osseotite Certain Tapered Group C
  Interventions: Device: Osseotite Certain Tapered Group C

INTERVENTIONS:
Device: Osseotite Certain Tapered Group A — Osseotite Certain Tapered with different surface roughness
  Other Names: Osseotite endosseous dental implant
  Arms: Roughness group A
Device: Osseotite Certain Tapered Group B — Osseotite Certain Tapered with different surface roughness
  Other Names: Osseotite endosseous dental implant
  Arms: Roughness Group B
Device: Osseotite Certain Tapered Group C — Osseotite Certain Tapered with different surface roughness
  Other Names: osseotite endosseous dental implant
  Arms: Roughness Group C

SUMMARY:
A study where dental implants with different roughened surfaces will be evaluated for the ability to resist countertorque forces.

DETAILED DESCRIPTION:
This study on dental implants with different roughened surfaces will assess its ability to resist countertorque testing at various study time points and demonstrate high success

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and older than 18 years of age
* patients needing at least one dental implant to treat partial edentulism
* patients physically able to tolerate surgical and restorative dental procedures
* patients agreeing to all protocol visits

Exclusion Criteria:

* patients with infection or severe inflammation at the intended treatment sites
* patients smoking greater than 10 cigarettes per day
* patients with uncontrolled diabetes mellitus
* patients with uncontrolled metabolic diseases
* patients who received radiation treatment to the head in the past 12 months
* patients needing bone grafting at the intended treatment sites
* patients known to be pregnant at screening visit
* patients with para-functional habits like bruxing and clenching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Primary stability countertorque measures | 6 weeks
  Resistance to countertorque measures showing primary stability and success of the implant

SECONDARY OUTCOMES:
Cumulative success rate | 2 years
  Crestal bone regression (amount of bone loss measured) and equivalence in integration success (implant mobility)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Acuna, DDS, Principal Investigator — Hospital San Jose
Locations (1):
- Hospital San Jose, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No